CLINICAL TRIAL: NCT02411890
Title: The Comparison of Postoperative Analgesia Between Adductor Canal Block and Femoral Nerve Block After Arthroscopic ACL Reconstruction With Hamstring Graft: A Randomized Controlled Trial
Brief Title: Postoperative Pain Between ACB and FNB After ACLR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Thammasat University (Other)
Responsible Party: Principal Investigator, Alisa Seangleulur, Department of Anesthesiology, Thammasat University, Thammasat University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MTU-EC-AN-6-014/58
Record Dates: First submitted 2015-03-29; First posted 2015-04-08 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Pain, Postoperative; Knee Arthroscopy; Anterior Cruciate Ligament/Surgery
Keywords: postoperative pain; femoral nerve block; adductor canal block; anterior cruciate ligament reconstruction
MeSH Terms: conditions — Pain, Postoperative | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adductor canal block (Experimental): Adductor canal block (active) + Femoral nerve block (sham block)
  Interventions: Procedure: Adductor canal block (active); Procedure: Femoral nerve block (sham block)
- Femoral nerve block (Active Comparator): Femoral nerve block (active) + Adductor canal block (sham block)
  Interventions: Procedure: Femoral nerve block (active); Procedure: Adductor canal block (sham block)

INTERVENTIONS:
Procedure: Adductor canal block (active) — adductor canal block: single injection, 0.5% levobupivacaine 15 ml with adrenaline 5 µg/ml, ultrasound guidance with nerve stimulator
  Arms: Adductor canal block
Procedure: Femoral nerve block (active) — femoral nerve block: single injection, 0.25% levobupivacaine 30 ml with adrenaline 5 µg/ml, ultrasound guidance with nerve stimulator
  Arms: Femoral nerve block
Procedure: Femoral nerve block (sham block) — 30 mL of normal saline injected into absorbing cloth through stump needle at the inguinal area but not penetrating skin, ultrasound guidance and nerve stimulator with percutaneous electronic guidance to create quadriceps contraction before injection
  Arms: Adductor canal block
Procedure: Adductor canal block (sham block) — 30 mL of normal saline injected into absorbing cloth through stump needle at the midfemoral area but not penetrating skin, ultrasound guidance and nerve stimulator with percutaneous electronic guidance without muscle contraction
  Arms: Femoral nerve block

SUMMARY:
The aim of this study is to compare the efficacy in pain relief within 24 hours between adductor canal block and femoral nerve block after anterior cruciate ligament reconstruction with hamstring graft.

DETAILED DESCRIPTION:
After approval from institutional ethic committees, Thammasat University Hospital, patients who meet the eligible criteria will be asked for informed consent. Randomization will be performed by computerization with varied block sizes (4 and 6), and the sequence of randomization will be concealed by sealed envelopes. Once given informed consent, the investigator opened the sealed envelope, which randomized the patient to the adductor canal block group (ACB), or the femoral nerve block group (FNB).

The day before surgery day, patients who meet the eligible criteria will ask for the informed consent from blinded research assistant. They will obtain patients' demographic data, preoperative pain scores, and quadriceps strength. They will be recommended how to evaluate pain score and use the patient-controlled analgesia.

In the block room, patients will be sedated with midazolam 2-3 mg intravenously. The nerve block will be performed before spinal anesthesia by unblinded anesthesiologists. During block, the patients will be blinded by sham block. In ACB group, patients will receive sham block of femoral nerve at inguinal area, and then ACB will be performed, while in FNB group, patients will receive FNB, and then sham block will be performed in the mid-femoral area.

After standard monitored, the saphenous nerve will be blocked in the ACB group under ultrasound guidance using linear probe (9 mHz, GE Healthcare®) with nerve stimulator (Payunk®) at midfemoral level. When the needle tip is positioned, the nerve stimulator is turned on and set to deliver a current of 0.5 mA at a frequency of 2 Hz and pulse duration of 0.1 ms. The presence of a quadriceps muscle twitch, if elicited, will be recorded, and the needle was re-positioned until the muscle twitch disappeared. Then, 0.5% levobupivacaine with adrenaline 5 µg/ml 15 ml will be injected.

The femoral nerve block is also performed in the FNB group under ultrasound guidance using linear probe (9 mHz, GE Healthcare®) and nerve stimulator (Payunk®). With ultrasound guidance, the femoral nerve is identified in femoral triangle near to femoral artery, and when the needle tip is in proper position in the ultrasound image, the nerve stimulator is used to confirm, the presence of quadriceps twitching at the current less than 0.5 mA, and the absence of quadriceps twitching at the current more than 0.2 mA. After that, 30 ml of 0.25% levobupivacaine with adrenaline 5 µg/ml is injected.

During performing both blocks, patients' eyes will be closed. The sham block involves an ultrasound survey at inguinal area in ACB group and mid-femoral area in FNB group, stump needle is marked at the injection site but not penetrating skin. 10 or 30 mL of saline depending on type of sham block will be injected into an absorbing cloth. Opaque plaster will be used for both block sites.

Fifteen minutes after ACB or FNB, the success of block is evaluated by blinded investigators. Loss of sensation at the either infrapatellar region or medial of calf will be tested every 5 mins. Fail block is documented, if there is no loss of sensation greater than 30 mins after block performed. Then, spinal anesthesia is performed with 0.5% isobaric or heavy marcaine 2.5-3.5 ml.

In the operative room, patients will receive cefazolin 1 gm, and ketorolac 30 mg intravenously before skin incision. Tourniquet 350 mmHg will be applied on operated thigh and limited time is no longer than 120 mins. Drain will be inserted, and knee brace or Jone's bandage will be applied postoperatively in all patients.

Postoperatively, all patients received disposable patient-controlled analgesia (PCA) for parenteral morphine as needed to control VAS less than 4 with setting PCA dose 2.5 mg (patients ≤ 60 years) 2 mg (patients ≥ 60 years), no basal rate, lock out 5 mins. Postoperative analgesic regimen are ketorolac 30 mg IV 8 hours after intraoperative dose, Etoricoxib (90) 1 tab oral once daily, paracetamol (500) 1 tab oral every 6 hours, reparil 2 tab oral tid, and myonal 1 tab oral tid. Drain will be removed in postoperative day 1 by surgeons and patients will be allowed to walk with crutches after drain removes Outcomes The primary outcome is VAS at 24 hours during activity . The patients will be instructed in the use of the 0 to 100 mm visual analogue scale (VAS) with 0 and 100 mm referring to 'no pain' and 'worst pain imaginable', respectively, at inclusion to the study.

VAS also assessed at 4 hour after surgery and then every 4 hours, at rest, and activity until 24 hours.

Total opioid consumption in first 24 hours and first time that patient pressing PCA is also recorded. Opioid side effects (nausea vomiting, pruritus, respiratory depression, urinary retention) will be recorded. Nausea vomiting, and pruritus will be recorded as 0-2 scales: 0=none, 1=mild symptom but no need treatment, 2=severe symptom and need medical treatment). Respiratory depression will be recorded as yes (respiratory rate≤8 per minute), and no. Urinary retention will be measured as yes (need urinary catheterization), and no.

Quadriceps strength will be assessed as maximum voluntary isometric contraction (MVIC) preoperatively, 8-12, and 24 hours postoperatively with handheld dynamometer (HHD, Lafayette Instrument, Lafayette, IN) which has been already calibrated. The strength will be evaluated by blinded research assistant, and use the Velcro strap to fix the dynamometer to reduce interrater variability. The patients will sit with 60 degree knee flexion, with attach the HHD at 5 cm above transmalleolar axis. The patients will be asked for extend their knee as forcefully as possible in 3 seconds with the instruction of the assessors (push-push-push-pause). The strength will be measured for 3 times and the maximum value will be used. Then, the maximal torque will be calculated by multiplying the maximal force (newtons) with the distance between femoral condyle and HHD (meters). After each contraction, the level of pain is quantified with use of a 0-100 point VAS.

Timing for readiness for hospital discharge within 24 hours will also be recorded. The criteria of readiness hospital discharge is patient is alert and responsive to questioning, show acceptable pain and nausea control, able to urinate, able to walk with crutches. The actual time of discharge and the reason of delayed discharge will also be recorded. All outcomes are assessed by blinded outcome assessors, who do not involved in other parts of this study.

Statistical analysis Continuous data will be presented as mean (SD) or median (IQR) as appropriate, and categorical data will be presented as frequency (percentage).The comparison between continuous data will be performed by t-test or Mann-Whitney U test depending on the distribution of data. Pain scores in first 24 hours were compared after calculating the area under the curve for the interval 2 to 24 hours.Categorical variables will be compared by chi-square or Fischer-exact test. P values less than 0.05 shows statistical significance. Statistical analysis will be performed by using STATA (13.0) software.

ELIGIBILITY:
Inclusion Criteria:

* arthroscopic anterior cruciate ligament reconstruction with hamstring graft at Thammasat University Hospital.
* age 15-80 years
* ASA class I-III

Exclusion Criteria:

* refuse to participate the study
* morbid obesity (BMI ≥ 35 kg.m2)
* allergic to any medication in the study
* chronic opioid use or abuse
* lower extremity neurological dysfunction
* patients who cannot cooperate and assess pain score themselves.

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Pain score (VAS) during activity | 24 hours postoperative
  Pain score during activity measured on Visual Analog Scale postoperative 24 hours. Adductor canal block VS Femoral nerve block

SECONDARY OUTCOMES:
Opioid consumption | 0-24 hours postoperative
  Intravenous morphine consumption (milligrams) during 0-24 hours from patient controlled analgesia. Adductor canal block vs Femoral nerve blockanalgesia.
Pain score (VAS) at rest | 4, 8, 12, 16, 20, 24 hours postoperative
  Adductor canal block vs Femoral nerve block
Pain score (VAS) at activity | 4, 8, 12, 16, 20 hours postoperative, and during quadriceps strength testing
  Adductor canal block vs Femoral nerve block
duration (hours) after surgery-first time that patients pressing PCA | 0-24 hours postoperative
  Adductor canal block vs Femoral nerve block
The reduction of quadriceps strength from preoperative period both knees | 8-12, 24 hours
  Quadriceps strength measured on the maximum voluntary isometric contraction with hand-held dynamometer. Adductor canal block vs Femoral nerve block
Postoperative nausea and vomiting | 0-24 hours postoperative
  Rating scale 0-2. Adductor canal block vs Femoral nerve block
Postoperative pruritus or rash | 0-24 hours postoperative
  Rating scale 0-2. Adductor canal block vs Femoral nerve block
Postoperative urinary retention | 0-24 hours postoperative
  Dichotomous outcome (Yes/No). Adductor canal block vs Femoral nerve block
Postoperative respiratory depression | 0-24 hours postoperative
  Dichotomous outcome (Yes/No). Adductor canal block vs Femoral nerve block

CONTACTS AND LOCATIONS:
Overall Officials: Alisa Seangleulur, MD, Principal Investigator — Thammasat University
Locations (1):
- Thammasat University Hospital, Khlong Luang, Changwat Pathum Thani, Thailand

REFERENCES:
- [Result] Beck PR, Nho SJ, Balin J, Badrinath SK, Bush-Joseph CA, Bach BR Jr, Hayden JK. Postoperative pain management after anterior cruciate ligament reconstruction. J Knee Surg. 2004 Jan;17(1):18-23. doi: 10.1055/s-0030-1247142. PMID 14971669
- [Result] Chisholm MF, Bang H, Maalouf DB, Marcello D, Lotano MA, Marx RG, Liguori GA, Zayas VM, Gordon MA, Jacobs J, YaDeau JT. Postoperative Analgesia with Saphenous Block Appears Equivalent to Femoral Nerve Block in ACL Reconstruction. HSS J. 2014 Oct;10(3):245-51. doi: 10.1007/s11420-014-9392-x. Epub 2014 Jun 7. PMID 25264441
- [Result] Hanson NA, Derby RE, Auyong DB, Salinas FV, Delucca C, Nagy R, Yu Z, Slee AE. Ultrasound-guided adductor canal block for arthroscopic medial meniscectomy: a randomized, double-blind trial. Can J Anaesth. 2013 Sep;60(9):874-80. doi: 10.1007/s12630-013-9992-9. Epub 2013 Jul 3. PMID 23820968